CLINICAL TRIAL: NCT00210301
Title: Combination Therapy (Provigil + Avonex) in the Treatment of Attention Problems in Patients With Relapsing-Remitting MS
Brief Title: Combination Therapy (Provigil + Avonex) to Treat Cognitive Problems in MS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute for Clinical Research (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2006-09-07 (Estimated); Status verified 2005-08

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: MS; cognition; attention; fatigue
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Fatigue | interventions — Modafinil

INTERVENTIONS:
Drug: Provigil (modafinil)

SUMMARY:
MS has been associated with fatigue, attention problems, and a number of cognitive difficulties. There is no treatment approved yet to treat these problems. We hypothesize that the addition of Provigil to an existing immunomodulatory agent (Avonex) will lead to improved fatigue, attention, and overall cognition in MS patients with attention problems.

DETAILED DESCRIPTION:
MS has been associated with fatigue, attention problems, and a number of cognitive difficulties. There is no treatment approved yet to treat these problems. Although certain immunomodulatory treatments may slow the progression of cogntiive difficulties, they are not therapy for the progression of or new onset of such problems. Therefore, in order to treat such problems, it is likely that adjunctive medications focused on fatigue and cognition are needed. We hypothesize that the addition of Provigil to an existing immunomodulatory agent (Avonex) will lead to improved fatigue, attention, and overall cognition in MS patients with attention problems.

Study Period: 6 to 12-month competitive enrollment period, two groups (Avonex and Avonex +Provigil 200 mg QD ) undergo baseline (prior to starting Provigil), 2-month, and 4-month neuropsychological evaluations. Total length of study, once initiated, (including 2 month preparation period, 6 to 12-month competitive enrollment period through final four-month visit) is 12 to 18 months.

Primary Objective: To investigate whether Provigil in combination with Avonex is safe, and tolerable in patients with RRMS.

Secondary Objectives:

1. To determine whether Provigil (modafinil) in combination with Avonex(interferon β-1a) is useful in treating deficits in attention, as measured by objective neuropsychological tests, in patients with RR-MS
2. To determine whether combination therapy (Avonex +Provigil) favorably impacts other domains of cognition that are reliant on attention (e.g., memory, psychomotor functioning), as measured by objective neuropsychological tests, in patients with RR-MS
3. To determine whether improvement in fatigue (related to treatment) predicts improvements in attention and cognitive performance in MS patients

ELIGIBILITY:
Inclusion Criteria:

* Patients entering the study will:

  * Be taking Avonex
  * Have normal laboratory blood tests and EKG
  * Be complaining of attention problems to treating neurologist
  * Be English-speaking males and females between the ages of 25 and 60, inclusive [If patient is female, she must

    * Be surgically sterile; or
    * Be 2 years postmenopausal; or
    * If of child-bearing potential, must be using a medically accepted method of birth control and agree to continue to use this method for the duration of the study (i.e., barrier method with spermicide, steroidal contraceptive [oral, implanted, and Depo-Provera contraceptives must be used in conjunction with a barrier method], IUD, or abstinence)]
  * Have clinically definite RR MS with disease duration of less than 10 years
  * Have an EDSS score between 0 and 5.5
  * Have corrected vision of no worse than 20/50
  * Have between 10 and 20 years of education
  * Be cerebral-stimulant free for at least one week prior to Attention Screening
  * Be able to complete self-rating scales and cognitive assessment tools
  * Have provided written informed consent
  * To have performed at least one standard deviation below normative expectation on at least two of four measures in the attention screening evaluation

Exclusion Criteria:

* Patients entering the study will NOT:

  * A history of heart disease or liver dysfunction
  * Have abnormal EKG or laboratory blood work,
  * Have a history of psychosis
  * Be a significant risk of suicide
  * Be abusing alcohol (current and within last 2 years)
  * Be abusing controlled substances (current and within last 2 years)
  * Have any medical ailment which can produce fatigue, such as lupus, anemia or thyroid disease
  * Have any history of clinical deviation from normal ranges in the physical examination
  * Have an unstable medical disorder, or medical contraindication to the use of Provigil
  * Have any history of head injury, seizures, or neurological conditions involving the central nervous system other than RR MS
  * Have any disorder that may interfere with drug absorption, distribution, metabolism, or excretion, including gastrointestinal surgery
  * Be a pregnant or lactating female (any patient becoming pregnant during the study will be discontinued)
  * Have received any investigational product within 30 days of Cognitive Screening
  * Have upper extremity dysfunction that prohibits them from using a computer mouse writing with a pencil
  * Be colorblind

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-01

PRIMARY OUTCOMES:
Comparison of AE's and SAE's to determine safety of combination

SECONDARY OUTCOMES:
Full neuropsychological test battery (including fatigue measures) to assess effect on fatigue and cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Wilken, Ph.D., Principal Investigator — Institute for Clinical Research
Locations (1):
- Veterans Affairs Medical Center, Washington D.C., District of Columbia, United States